CLINICAL TRIAL: NCT06357468
Title: Analysis of Pain Management and Pain Perception Intrapartum and Postpartum in Women with Vaginal Births in Difference Between Physician-led and Midwife-led Birth
Status: Completed | Type: Observational
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Marcus Riemer, MD, Principal Investigator, Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: UKGEB003
Record Dates: First submitted 2024-03-30; First posted 2024-04-10 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Pain, Labor
MeSH Terms: conditions — Labor Pain | interventions — Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- physician-led births
  Interventions: Other: midwife-led births in low risk women in pregnancy
- midwife-led births

INTERVENTIONS:
Other: midwife-led births in low risk women in pregnancy — Pregnant women in the low-risk collective are cared for in a midwife-led delivery room if they wish to have a natural birth
  Groups: physician-led births

SUMMARY:
The aim of the analysis is to describe the differences and similarities in obstetric pain management and pain perception intrapartum and postpartum in women with vaginal births in contrast to physician-led births and midwife-led births

ELIGIBILITY:
Inclusion Criteria:

* Understanding written and spoken German
* Declaration of consent

Exclusion Criteria:

* under 18 years
* incomplete answered questionaire

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pregnant women under birth
Sampling Method: Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pain perception | intrapartum (start of labour until end of labour) and postpartum first 3 days after birth
  Measured by visual pain scale (1-10)

SECONDARY OUTCOMES:
Satisfaction with pain therapy | intrapartum (start of labour until end of labour) and postpartum first 3 days after birth
  Measured by visual analog scale (1-10)
Pain perception in women with perineal tear grade III | postpartum first 3 days after birth
  Measured by visual pain scale (1-10)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Halle, Halle, Saxony-Anhalt, Germany

IPD SHARING:
Plan to Share IPD: No